CLINICAL TRIAL: NCT05939713
Title: A Multi-center, Single Arm, Real-World Registry Assessing the Clinical Use of the Cera™ VSD Occluder
Brief Title: Cera™ VSD Occluder Post Market Clinical Follow-up
Status: Completed | Type: Observational
Sponsor: Cardiac Children's Foundation Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: LT/TS/29I-01N-01
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Ventricular Septal Defect
Keywords: Cera VSD occluder; Observational; Retrospective; Multi-center
MeSH Terms: conditions — Heart Septal Defects, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- VSD subjects: Patients with a confirmed diagnosis of Ventricular Septal Defect (VSD) and implanted with the Cera VSD occluder as per IFU instructions
  Interventions: Device: Cera™ VSD occluder implantation

INTERVENTIONS:
Device: Cera™ VSD occluder implantation — To collect data from patients who have implanted with the device before 2022.

SUMMARY:
The objective of this post-market registry is to assess the safety and performance of the Lifetech Cera™ VSD occluder in a real-world and on-label fashion.

DETAILED DESCRIPTION:
The study intends to collect data from patients who have implanted with the device before 2022. The study is expected to completed by the end of 2024.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of Ventricular Septal Defect (VSD) and implanted with the investigational device as per IFU instructions

Exclusion Criteria:

* Patients did not conduct any follow up visit after hospital discharge.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study intends to collect data from patients who have implanted with the device before 2022
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Procedural success | 6 months post-implantation
  Defined as a composite of:
  1. Absence of complete atrioventricular block (third degree AV block) needing pacemaker implantation, device embolization, severe aortic regurgitation requiring surgical repair or device or procedure related death, assessed at 6 months post-implantation.
  2. Successful closure of the defects, with no, trivial or small residual shunt confirmed by Doppler echocardiography at 6 months post-implantation .

SECONDARY OUTCOMES:
Incidence of moderate or large residual shunt | at procedure, 6 months and 12 months post-implantation
Incidence of new onset complete AV block (third-degree AV block) or any new onset arrhythmia needing for pacemaker implantation, or new onset left bundle branch block (LBBB); | from attempted procedure to 24 months post-implantation
Incidence of new onset second-degree AV block | from attempted procedure to 24 months post-implantation
Incidence of new onset severe aortic or tricuspid regurgitation | from attempted procedure to 24 months post-implantation
Incidence of device-related thrombosis (DRT) | from attempted procedure to 24 months post-implantation
Incidence of device embolization | from attempted procedure to 24 months post-implantation
Incidence of device or procedure related Adverse Events (AEs) | from attempted procedure to 24 months post-implantation
Incidence of device or procedure related Serious Adverse Events (SAEs) | from attempted procedure to 24 months post-implantation
Incidence of Device Deficiencies (DD) | from attempted procedure to 24 months post-implantation
Incidence of death | from attempted procedure to 24 months post-implantation

CONTACTS AND LOCATIONS:
Overall Officials: Jou-Kou Wang, Principal Investigator — National Taiwan University Hospital
Locations (8):
- Taiwan (8):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang-Gung Memorial Hospita, Taoyuan District

IPD SHARING:
Plan to Share IPD: No